CLINICAL TRIAL: NCT04451447
Title: Effectiveness and Sensitivity of White Test Versus Conventional Saline Test in Minimizing Biliary Leak in Partial Liver Resection in Living Donor Liver Transplant
Brief Title: White Test in Intra-operative Detection of Donor Biliary Leak in LDLTx.
Acronym: LDLTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amr Abdelaal (Other)
Responsible Party: Sponsor-Investigator, Amr Abdelaal, professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: White test in LDLTx
Record Dates: First submitted 2020-06-27; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Bile Leak
Keywords: White test, Donor, liver transplantation, living donor
MeSH Terms: interventions — SMOFlipid

STUDY DESIGN:
Intervention Model Description: Non randomized controlled Interventional trial Compare the study group with a historical cohort.
Who Masked: Outcomes Assessor
Masking Description: Compare one group with a historical cohort. masked outcome for the tested and control arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- white test arm (Experimental): The White test uses fat emulsion (SMOFLIPID), which is a lipid emulsion with a lipid content of 0.2 grams/mL in 100 mL, 250 mL, and 500 Ml that is normally used for parenteral nutrition, for localization of bile leakage.
  Interventions: Procedure: The White test uses fat emulsion (SMOFLIPID), for localization of bile leakage.
- Saline test arm (Other): The conventional intra-operative saline test, which involves injecting an isotonic sodium chloride solution through the cystic duct, has been used for detection of leaking points from the transected liver surface.
  Interventions: Procedure: Saline test (routine test)

INTERVENTIONS:
Procedure: The White test uses fat emulsion (SMOFLIPID), for localization of bile leakage. — The White test uses fat emulsion (SMOFLIPID), which is a lipid emulsion with a lipid content of 0.2 grams/mL in 100 mL, 250 mL, and 500 Ml that is normally used for parenteral nutrition, for localization of bile leakage.
  Arms: white test arm
Procedure: Saline test (routine test) — The conventional intra-operative saline test, which involves injecting an isotonic sodium chloride solution through the cystic duct, has been used for detection of leaking points from the transected liver surface.
  Arms: Saline test arm

SUMMARY:
Biliary leak is a common complication after partial liver resection in living donor liver transplant. It debases the quality of the postoperative course and affects morbidity and mortality. Detecting and localizing sites of biliary leak intraoperatively through bile leakage testing is important as it helps in detection of bile leaking points on the cut surface and decrease post-operative bile leak.

In this study we will assess the efficacy and sensitivity of using White test in comparison to conventional saline test in detecting intra operative bile leakage in liver donor.

The White test uses fat emulsion (SMOFLIPID), which is a lipid emulsion with a lipid content of 0.2 grams/mL in 100 mL, 250 mL, and 500 Ml that is normally used for parenteral nutrition, for localization of bile leakage. The use of fat emulsion in bile leakage tests does not require special equipment, contaminate the wound, cause allergic reaction or damage the bile duct and surrounding tissues.

DETAILED DESCRIPTION:
Postoperative bile leakage is one of the commonest causes of sepsis and liver failure after liver resection in liver donor [ Yamashita YI et al, 2001 ] [ Langer D et al, 2011 ].Various studies have showed that the incidence of postoperative bile leakage after liver resection ranges from 3 to 27% [ Erdogan D et al, 2008 ] [ Ishii H et al, 2011 ].

The timely detection and repair of intraoperative bile leakage is extremely important, but small leakage points are often difficult to detect [ Liu Z et al, 2012 ]. There are different methods for detecting and or preventing bile leakage after partial liver resection, including bile leakage tests, which detect open bile duct stumps on the resection surface through increasing fluid pressure within the duct [ Lo CM et al, 1998 ].

The conventional intraoperative saline test, which involves injecting an isotonic sodium chloride solution through the cystic duct, has been used for detection of leaking points from the transected liver surface [ Ijichi M et al, 2000 ]. One of the main problems in using the conventional bile leakage test is that the isotonic sodium chloride solution is a transparent solution. Therefore, it is hard to detect the point of bile leakage. A previous randomized study stated that there is no advantage to using the isotonic sodium chloride solution for the bile leakage test during liver resection [ Ijichi M et al, 2000 ].

During the past decade, several bile leak tests have been proposed, with none gaining wide acceptance. The intraductal injection of saline is a low-cost and reproducible technique, but the transparent solution makes this technique inadequate for detecting small ducts. The injection of dye solutions (e.g. methylene blue and indocyanine green) has been recommended. However, these solutions need to be dense in order to allow the visualization of the leak site. The related disadvantages of this approach include the following: 1) the indelible coloration of the transection surface, which can mask additional small open ducts, 2) the impossibility to wash out the staining and, consequently, 3) potential reduced sensitivity for the detection of leak with repeated tests. Some centres have reported the saturation of the cut surface of the liver with hydrogen peroxide to detect bile leaks, however this practice comes with a potential risk of expansion air embolism via open hepatic veins.

The White test uses fat emulsion (SMOFLIPID), which is a lipid emulsion with a lipid content of 0.2 grams/mL in 100 mL, 250 mL, and 500 Ml that is normally used for parenteral nutrition, for localization of bile leakage (Morris-Stiff G et al., 2009). The use of fat emulsion in bile leakage tests does not require special equipment, contaminate the wound, cause allergic reaction or damage the bile duct and surrounding tissues. It can easily be repeated the number of times necessary to detect and close all leakage points, can pinpoint even small leaks and is inexpensive. This technique is easier to perform than fluorescent imaging, and is more sensitive and reliable compared with saline bile leakage test used alone (Leelawat K et al., 2012; Kaibori M et al., 2011).

Recently, intraoperative application of the White test has been demonstrated to reduce the incidence of postoperative bile leakage [ Li J et al, 2009 ] [ Nadalin S et al, 2008 ]. In this technique, bile leakage sites on the transected liver surface are noted by injecting a fat emulsion solution through the cystic duct. The previous prospective observational studies suggested that the fat emulsion solution used in the White test is easily recognized, innocuous and harmeless to the tissues, and can be easily removed without misleading tissue staining [ Li J et al, 2009 ] [ Nadalin S et al, 2008 ]. Therefore, this prospective study will assess whether the White test is better than the conventional saline test for the intraoperative detection of bile leakage and better prevention of post-operative bile leakage in partial resection in living donor liver transplant.

ELIGIBILITY:
Inclusion Criteria:patients who are candidate for liver donation) Criteria for donor of living donor liver transplantation):

1. Potential donors must be healthy volunteers between the ages of 18 and 45 years.
2. BMI must be up to 28.
3. Blood group must be compatible; Rh compatibility was not a significant criterion.
4. Donors should have normal liver function and no medical comorbidities.
5. Liver biopsy was done to ensure that there is no occult hepatic pathology and to establish the degree of steatosis that should be less than 20%.
6. Donors must have no history of upper abdominal surgery.

Exclusion Criteria:

Intra operative vascular or biliary complication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Intra-operative detection of bile leak points | Immediate Intra-operative
  Detection and suturing of bile leak points

SECONDARY OUTCOMES:
post-operative bile leak | Early post-operative (one month)
  post-operative bile leak - Biloma
Surgical site infection | Early post-operative (one month)
  Infected biloma

CONTACTS AND LOCATIONS:
Overall Officials: amr abdelaal, prof, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No